CLINICAL TRIAL: NCT04933240
Title: Tamoxifen Versus Estradiol in the Prevention of Unscheduled Bleeding in Etonogestrel Implant Users, a Randomized Controlled Pilot Trial
Brief Title: Tamoxifen Versus Estradiol for Unscheduled Bleeding in Etonogestrel Implant Users, a Randomized Pilot Trial
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Anticipated funding was not received
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HM20021901
Record Dates: First submitted 2021-06-14; First posted 2021-06-21 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Vaginal Bleeding
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Tamoxifen; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tamoxifen (Active Comparator): tamoxifen 10mg daily for 7 days
  Interventions: Drug: Tamoxifen Citrate 10Mg Tab
- Estradiol (Active Comparator): estradiol 1mg daily for 7 days
  Interventions: Drug: Estradiol
- placebo (Placebo Comparator): placebo daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamoxifen Citrate 10Mg Tab — nonsteroidal antiestrogen for oral administration in 10 mg tablets. Each tablet contains 15.2 mg of tamoxifen citrate which is equivalent to 10 mg of tamoxifen.
  Other Names: NOLVADEX
  Arms: Tamoxifen
Drug: Estradiol — estradiol tablets for oral administration contains 1 mg of micronized estradiol per tablet.
  Other Names: ESTRACE
  Arms: Estradiol
Drug: Placebo — A sugar tablet that does not contain any active medicine
  Other Names: Inactive drug
  Arms: placebo

SUMMARY:
The purpose of this research study is to evaluate the ability of medicines called tamoxifen or estradiol to prevent annoying vaginal bleeding for arm implant users.

DETAILED DESCRIPTION:
This pilot study compares the use of tamoxifen to estradiol to placebo for seven days once a month up to 5 months in contraceptive implant users starting from the time of implant initiation. Participants will record bleeding and satisfaction response in a daily text diary.

ELIGIBILITY:
Inclusion Criteria:

* etonogestrel implant users
* at time of and/or within 21 days of initial use of etonogestrel implant placement
* must agree not to take additional hormonal therapy during the study trial period

Exclusion Criteria:

* within 6 months following vaginal or cesarean delivery
* within 6 weeks following abortion
* currently breastfeeding
* positive pregnancy test
* contraindications to tamoxifen or estrogen
* history of thromboembolism
* undiagnosed abnormal uterine bleeding
* active cervicitis
* bleeding disorder
* use of anticoagulation medications
* an unwillingness or inability to keep a daily menstrual diary or to follow the study criteria

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Duration of bleeding free days | Up to 28 days
  Number of days of no spotting or bleeding after initiation of first treatment until day of subsequent bleeding

SECONDARY OUTCOMES:
Total number of bleeding free days | Up to 24 weeks
  Total number of no spotting or bleeding days
Days to first re-treatment | Up to 24 weeks
  Number of days between first and second use of medication
Total number of re-treatments | Up to 24 weeks
  Total number of times participant used treatment medication
Satisfaction with bleeding | Up to 24 weeks
  Average satisfaction with bleeding will be assess using daily text surveys. Participants will rate degree of satisfaction with bleeding with the use of symbols (emojis): 1) completely unsatisfied, 2) somewhat unsatisfied, 3) neutral, 4) somewhat satisfied, 5) completely satisfied.
Affects on daily life activities | Up to 24 weeks
  The average affect of bleeding on daily life activities will be assess using daily text surveys. Participants will rate the degree of affects of bleeding on daily life with the use of a visual analogue scale from 0 (no affects) to 100 (highest possible affects)

CONTACTS AND LOCATIONS:
Overall Officials: Frances Casey, MD, MPH, Principal Investigator — VCU Health System
Locations (2):
- United States (2):
  - Shanthi Ramesh, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mansour D, Fraser IS, Edelman A, Vieira CS, Kaunitz AM, Korver T, Pong A, Lin J, Shah AK, Fox M, Rekers H, Creinin MD. Can initial vaginal bleeding patterns in etonogestrel implant users predict subsequent bleeding in the first 2 years of use? Contraception. 2019 Oct;100(4):264-268. doi: 10.1016/j.contraception.2019.05.017. Epub 2019 Jun 6. PMID 31176688
- [Background] Edelman AB, Kaneshiro B, Simmons KB, Hauschildt JL, Bond K, Boniface ER, Jensen JT. Treatment of Unfavorable Bleeding Patterns in Contraceptive Implant Users: A Randomized Controlled Trial. Obstet Gynecol. 2020 Aug;136(2):323-332. doi: 10.1097/AOG.0000000000003896. PMID 32649493
- [Background] Abdel-Aleem H, d'Arcangues C, Vogelsong KM, Gaffield ML, Gulmezoglu AM. Treatment of vaginal bleeding irregularities induced by progestin only contraceptives. Cochrane Database Syst Rev. 2013 Oct 21;2013(10):CD003449. doi: 10.1002/14651858.CD003449.pub5. PMID 24146298
- [Background] Abdel-Aleem H, Shaaban OM, Amin AF, Abdel-Aleem AM. Tamoxifen treatment of bleeding irregularities associated with Norplant use. Contraception. 2005 Dec;72(6):432-7. doi: 10.1016/j.contraception.2005.05.015. Epub 2005 Aug 9. PMID 16307966
- [Background] DeCensi A, Puntoni M, Guerrieri-Gonzaga A, Caviglia S, Avino F, Cortesi L, Taverniti C, Pacquola MG, Falcini F, Gulisano M, Digennaro M, Cariello A, Cagossi K, Pinotti G, Lazzeroni M, Serrano D, Branchi D, Campora S, Petrera M, Buttiron Webber T, Boni L, Bonanni B. Randomized Placebo Controlled Trial of Low-Dose Tamoxifen to Prevent Local and Contralateral Recurrence in Breast Intraepithelial Neoplasia. J Clin Oncol. 2019 Jul 1;37(19):1629-1637. doi: 10.1200/JCO.18.01779. Epub 2019 Apr 11. PMID 30973790
- [Background] Buzdar AU, Hortobagyi GN, Frye D, Ho D, Booser DJ, Valero V, Holmes FA, Birmingham BK, Bui K, Yeh C, et al. Bioequivalence of 20-mg once-daily tamoxifen relative to 10-mg twice-daily tamoxifen regimens for breast cancer. J Clin Oncol. 1994 Jan;12(1):50-4. doi: 10.1200/JCO.1994.12.1.50. PMID 8270984
- [Background] Macpherson AM, Archer DF, Leslie S, Charnock-Jones DS, Makkink WK, Smith SK. The effect of etonogestrel on VEGF, oestrogen and progesterone receptor immunoreactivity and endothelial cell number in human endometrium. Hum Reprod. 1999 Dec;14(12):3080-7. doi: 10.1093/humrep/14.12.3080. PMID 10601100
- [Background] Leslie KK, Walter SA, Torkko K, Stephens JK, Thompson C, Singh M. Effect of tamoxifen on endometrial histology, hormone receptors, and cervical cytology: a prospective study with follow-up. Appl Immunohistochem Mol Morphol. 2007 Sep;15(3):284-93. doi: 10.1097/01.pai.0000213147.54901.12. PMID 17721273
- [Background] Archer DF, Philput CA, Weber ME. Management of irregular uterine bleeding and spotting associated with Norplant. Hum Reprod. 1996 Oct;11 Suppl 2:24-30. doi: 10.1093/humrep/11.suppl_2.24. PMID 8982742
- [Background] Thomas AM, Hickey M, Fraser IS. Disturbances of endometrial bleeding with hormone replacement therapy. Hum Reprod. 2000 Aug;15 Suppl 3:7-17. doi: 10.1093/humrep/15.suppl_3.7. PMID 11041216
- [Background] Alvarez-Sanchez F, Brache V, Thevenin F, Cochon L, Faundes A. Hormonal treatment for bleeding irregularities in Norplant implant users. Am J Obstet Gynecol. 1996 Mar;174(3):919-22. doi: 10.1016/s0002-9378(96)70326-5. PMID 8633669